CLINICAL TRIAL: NCT01259960
Title: Minimal Access Surgical Technique (MAST) in Obese Patients in Degenerative Lumbar Disease. A Prospective Long-term Evaluation.
Status: Completed | Type: Observational
Sponsor: Dr. Wolfgang Senker (Other)
Responsible Party: Sponsor-Investigator, Dr. Wolfgang Senker, Senior Consultant for orthopedy and orthopedic surgery, General Hospital Amstetten
Organization: General Hospital Amstetten (Other)
Other Study IDs: 2-Senker
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Degenerative Lumbar Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- BMI < 25: Body Mass Index (BMI) according to WHO definition. BMI < 25 is defined as 'normal weight'.
- 25 <= BMI < 30: Body Mass Index (BMI) according to WHO definition. BMI >= 25 and < 30 is defined as 'overweight'.
- BMI >= 30: Body Mass Index (BMI) according to WHO definition. BMI >= 30 is defined as 'obese'.

SUMMARY:
Being confronted more and more with obese as well as older patients, minimally invasive surgery is said to keep the surgical trauma low. The prospective long-term evaluation is the continuous monitoring of patients undergoing lumbar minimally invasive fusion surgery and analyzing the effect of body mass index (BMI) and wound healing.

ELIGIBILITY:
* All patients who will undergo minimally access surgical technique for degenerative lumbar disease fusion surger
* Patient willing to participate in observational study and who signs patient information and patient consent form
* patient older that 18 years
* all products will be used within intended use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who will undergo minimal access surgical technige for degenerative lumbar disease fusion
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2011-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Operation related complications | between operation and hospital discharge of patient
Post operative fever | between operation and hospital discharge of patient
Liquor leakage | between operation and hosital discharge of patient

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Senker, MD, Principal Investigator — General Hospital Amstetten
Locations (1):
- General Hospital, Amstetten, Austria